CLINICAL TRIAL: NCT04198428
Title: Clinic-Randomized Trial of Clinical Decision Support for Opioid Use Disorders in Medical Settings (COMPUTE 2.0)
Brief Title: Clinical Decision Support for Opioid Use Disorders in Medical Settings (COMPUTE 2.0)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry); Hennepin Healthcare Research Institute (Other); Geisinger Clinic (Other); Essentia Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CTN - 0095; UG1DA040316 (NIH)
Record Dates: First submitted 2019-12-03; First posted 2019-12-13 (Actual); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receives OUD-CDS (Experimental): Clinics will have access to the OUD-CDS (Opioid Wizard)
  Interventions: Other: Opioid Wizard
- Does not Receive the OUD-CDS (No Intervention): Clinics will not have access to the OUD-CDS (Opioid Wizard). These will be "usual care" clinics.

INTERVENTIONS:
Other: Opioid Wizard — The Opioid Wizard is an OUD clinical decision support tool for primary care providers to help assess, diagnose, and treat OUD in primary care (where appropriate).
  Arms: Receives OUD-CDS

SUMMARY:
Through CTN-0076-Ot (Clinical Decision Support for Opioid Use Disorders in Medical Settings: Pilot Usability Testing in an EMR (COMPUTE)), our team has iteratively developed and piloted a web-based and electronic health record (EHR)-integrated Opioid Use Disorder (OUD) Clinical Decision Support (CDS) system to offer expert guidance to primary care providers (PCPs) on the diagnosis and management of OUD. The OUD-CDS has been implemented within the EPIC EHR of one large care system and was piloted with 55 providers to ensure content validity and provider satisfaction. The team will now implement this OUD-CDS in a large multi-site clinic-randomized controlled trial to evaluate its impact on practice process measures and patient outcomes. The investigators also aim to prepare for scalability (i.e., integration into usual primary care practice after the study is complete) and dissemination by evaluating facilitators and barriers to implementation, determining the costs of implementation and maintenance, and assessing the short-term cost impacts of the OUD-CDS.

The study will include three large diverse care systems and randomize a minimum of 30 clinics to receive the OUD-CDS intervention or usual care (UC). In intervention clinics, the OUD-CDS will identify patients who are at high risk for OUD or diagnosed with OUD; use data stored in the EHR for each eligible patient to assemble treatment recommendations tailored to each patient's current needs; display these recommendations to PCPs via the OUD-CDS user interface; and store analytic data from all targeted visits. In UC clinics, the OUD-CDS will run invisibly in the background to identify high-risk or OUD patients, assemble treatment recommendations tailored to each eligible patient's needs, and store analytic data from all targeted visits.

DETAILED DESCRIPTION:
The proposed study will include 3 large diverse healthcare systems and randomize a minimum of 30 clinics equally within each system to receive the OUD-CDS intervention or UC. In intervention and UC clinics, the OUD-CDS will identify study-eligible patients, those who are at high risk for OUD or diagnosed with OUD; and will use data stored in the EHR to assemble treatment recommendations tailored to the needs of each study-eligible patient. In intervention clinics, these treatment recommendations will be displayed via the OUD-CDS user interface. Finally, data from all targeted visits in all randomized clinics will be stored in a data repository for analysis and reporting needs. The targeted visits for each study-eligible patient in all randomized clinics will be the index visit, the first visit at which the OUD-CDS identifies that the patient is study eligible, and all post-index visits through the end of the intervention period, regardless of continued eligibility. This pragmatic cluster-randomized design is the optimal design to effectively and efficiently implement this tool in primary care clinics while protecting against study contamination and allowing for collection of process and outcome data at UC clinics.

Mixed Methods Approach: Virtually every evidence-based intervention in medicine has turned out to be difficult to implement and maintain in real life practice and to fall far short of fidelity to the process used in randomized trials. As a result, a whole new field of dissemination and implementation research has been developing over the last 20 years. These studies have now gone well beyond the previous paradigm of focusing on changing the attitudes and behaviors of individual physicians to a growing awareness that the need instead is to alter the environment in which physicians work so that it is easier to do the desired evidence-based thing than to stick with old established habit patterns. That means focusing change efforts on organizational factors and practice systems. The Solberg conceptual framework has proven to be particularly helpful in clarifying this new approach.

Simultaneously, there has been increasing interest in transitioning effectiveness clinical trials from traditionally highly selective and controlled circumstances to pragmatic trials that make use of normal care delivery processes and patients.[35] The measurement of such trials has been facilitated by the development of a conceptual framework called RE-AIM, an acronym for 5 key facets of such studies - Reach, Effectiveness, Adoption, Implementation, and Maintenance. Recently, the developers of RE-AIM have recognized the need for more flexible use of this framework, greater use of qualitative methods to understand why interventions are not used consistently, and making adaptations in the implementation approach based on such understandings. The investigators propose to use the RE-AIM framework to guide (1) a monitoring system for intervention problems, (2) a mixed methods evaluation of the reasons for those problems, and (3) modification of the intervention to reduce those problems. These steps will be reiterated in a cyclic fashion, resulting in a more sophisticated approach to the long-standing quality improvement emphasis on Plan-Do-Study-Act rapid cycle tests of change. Furthermore, the team will take advantage of the staggered implementation of the study through three different care systems to ensure that the solutions for intervention problems in Site 1 are not assumed to be the same as the approach in subsequent sites without further RE-AIM monitoring and evaluation.

ELIGIBILITY:
Inclusion Criteria:

* be aged 18-75 years, inclusive, at the time of an index visit;
* have been diagnosed with OUD, currently prescribed MOUD, or identified by study algorithms as being at high risk of OUD.
* Be a patient at a study randomized clinic

Exclusion Criteria:

* those receiving active parenteral chemotherapy within the last year,
* those with stage 4 or equivalent cancer diagnosis
* those enrolled in hospice care or palliative care programs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10891 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Bart, MD PhD FACP DFASAM, Principal Investigator — Hennepin Healthcare; Rebecca Rossom, MD, MSCR, Principal Investigator — HealthPartners Institute
Locations (3):
- United States (3):
  - HealthPartners, Bloomington, Minnesota
  - Essentia Health, Duluth, Minnesota
  - Geisinger, Danville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rossom RC, Crain AL, Wright EA, Olson AW, Haller I, Haapala J, Dehmer SP, Hooker SA, Solberg L, O'Connor PJ, Borgert-Spaniol C, Gorodisher J, Miley K, Romagnoli K, Allen C, Tusing L, Ekstrom H, Appana D, Sperl-Hillen JM, Kobylinski M, Huntley K, McCormack J, Chen W, Bart G. Clinical Decision Support System for Primary Care of Opioid Use Disorder: A Randomized Clinical Trial. JAMA Intern Med. 2025 Sep 1;185(9):1079-1089. doi: 10.1001/jamainternmed.2025.2535. PMID 40658392
- [Derived] Olson AW, Bucaloiu A, Allen CI, Tusing LD, Henzler-Buckingham HA, Gregor CM, Freitag LA, Hooker SA, Rossom RC, Solberg LI, Wright EA, Haller IV, Romagnoli KM. 'Do they care?': a qualitative examination of patient perspectives on primary care clinician communication related to opioids in the USA. BMJ Open. 2025 Jan 7;15(1):e090462. doi: 10.1136/bmjopen-2024-090462. PMID 39773800
- [Derived] Olson AW, Haapala JL, Hooker SA, Solberg LI, Borgert-Spaniol CM, Romagnoli KM, Allen CI, Tusing LD, Wright EA, Haller IV, Rossom RC. The potential impact of clinical decision support on nonwaivered primary care clinicians' prescribing of buprenorphine. Health Aff Sch. 2023 Oct 11;1(4):qxad051. doi: 10.1093/haschl/qxad051. eCollection 2023 Oct. PMID 38756745

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: clinics
Period: Overall Study
Arm/Group | Receives OUD-CDS | Does Not Receive the OUD-CDS
Started | 5688; 46 clinics | 5509; 46 clinics
Completed | 5538; 46 clinics | 5353; 46 clinics
Not Completed | 150; 0 clinics | 156; 0 clinics
Not completed — Withdrawal by Subject | 150 | 156

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Receives OUD-CDS | Does Not Receive the OUD-CDS | Total
Number analyzed (Participants) | 5538 | 5353 | 10891
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (13.9) | 48.4 (13.9) | 48 (13.9)
Age, Customized [Count of Participants; unit: Participants]
  Age: 18-29 | 567 | 502 | 1069
  Age: 30-44 | 1877 | 1755 | 3632
  Age: 45-64 | 2387 | 2338 | 4725
  Age: 65-75 | 707 | 758 | 1465
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2979 | 2940 | 5919
  Male | 2559 | 2413 | 4972
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 186 | 145 | 331
  Not Hispanic or Latino | 5211 | 5149 | 10360
  Unknown or Not Reported | 141 | 59 | 200
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 246 | 122 | 368
  Asian | 34 | 18 | 52
  Native Hawaiian or Other Pacific Islander | 10 | 4 | 14
  Black or African American | 305 | 329 | 634
  White | 4697 | 4656 | 9353
  More than one race | 167 | 156 | 323
  Unknown or Not Reported | 79 | 68 | 147

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With OUD Diagnosis
Description: Patient has an ICD10 diagnosis code for OUD assigned at an encounter or added to the problem list
Time Frame: Index visit date through 30 days post-index, inclusive.
Population: Patients previously undiagnosed with OUD but identified as high risk by the OUD-CDS
Measure: Number; unit: participants
Arm/Group | Receives OUD-CDS | Does Not Receive the OUD-CDS
Number analyzed (Participants) | 2079 | 2074
participants | 36 | 24
Statistical Analysis 1: Comparison: Receives OUD-CDS vs Does Not Receive the OUD-CDS; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mixed-model regression adjusted for site and clinic factors balanced at randomization; Odds Ratio (OR) = 1.49

2. Primary Outcome: Number of Patients With Naloxone Rescue Kit Order
Description: Patient has a medication order for a naloxone rescue kit
Time Frame: Index visit date through 30 days post-index, inclusive.
Measure: Number; unit: participants
Arm/Group | Receives OUD-CDS | Does Not Receive the OUD-CDS
Number analyzed (Participants) | 5538 | 5353
participants | 80 | 40
Statistical Analysis 1: Comparison: Receives OUD-CDS vs Does Not Receive the OUD-CDS; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mixed-model regression adjusted for site and clinic factors balanced at randomization; Odds Ratio (OR) = 1.76

3. Primary Outcome: Number of Patients With a MOUD Order or Referral
Description: Patient has a medication order for a MOUD or referral for addiction treatment
Time Frame: Index visit date through 30 days post-index, inclusive.
Measure: Number; unit: participants
Arm/Group | Receives OUD-CDS | Does Not Receive the OUD-CDS
Number analyzed (Participants) | 5538 | 5353
participants | 785 | 517
Statistical Analysis 1: Comparison: Receives OUD-CDS vs Does Not Receive the OUD-CDS; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mixed-model regression adjusted for site and clinic factors balanced at randomization; Odds Ratio (OR) = 1.43

4. Primary Outcome: Days Covered by MOUD Prescription
Description: The sum of unique days covered by a MOUD order
Time Frame: Index visit date through 90 days post-index, inclusive, with 0 days assigned if there were no MOUD orders.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Receives OUD-CDS | Does Not Receive the OUD-CDS
Number analyzed (Participants) | 5538 | 5353
days | 84 [55 to 90] | 83 [55 to 90]
Statistical Analysis 1: Comparison: Receives OUD-CDS vs Does Not Receive the OUD-CDS; Test type: Superiority; p < 0.05, Mixed Models Analysis; Zero-inflated negative binomial mixed-model regression adjusted for site and clinic factors balanced at randomization; Risk Ratio (RR) = 0.99

5. Secondary Outcome: Emergency Department Visits Per Patient-year
Time Frame: pre: one year through one day prior to the index visit; post: index visit through one year post-index or date of death, whichever was first.
Measure: Number (95% Confidence Interval); unit: events per patient-year
Arm/Group | Receives OUD-CDS | Does Not Receive the OUD-CDS
Number analyzed (Participants) | 5538 | 5353
events per patient-year
  pre-index | 1.30 [1.11 to 1.52] | 1.37 [1.12 to 1.68]
  post-index | 1.06 [0.91 to 1.23] | 1.12 [0.97 to 1.47]
Statistical Analysis 1: Comparison: Receives OUD-CDS vs Does Not Receive the OUD-CDS; Test type: Superiority; p < 0.05, Mixed Models Analysis; Generalized estimating equation comparing post- to pre-index rates in OUD-CDS vs. Usual Care, adjusted for site and balancing factors; Risk Ratio (RR) = 0.93

6. Secondary Outcome: Hospitalizations Per Patient-year
Time Frame: as for outcome 5
Measure: Number (95% Confidence Interval); unit: events per patient-year
Arm/Group | Receives OUD-CDS | Does Not Receive the OUD-CDS
Number analyzed (Participants) | 5538 | 5353
events per patient-year
  pre-index | 0.40 [0.36 to 0.44] | 0.40 [0.35 to 0.46]
  post-index | 0.32 [0.29 to 0.36] | 0.33 [0.29 to 0.38]
Statistical Analysis 1: Comparison: Receives OUD-CDS vs Does Not Receive the OUD-CDS; Test type: Superiority; p < 0.05, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]; Risk Ratio (RR) = 1.01

7. Secondary Outcome: Healthcare Costs
Description: Healthcare costs for prescribed medications and clinical inpatient, emergency, and outpatient services incurred, as documented in insurance claims or clinical encounter data.
Time Frame: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: dollars
Arm/Group | Receives OUD-CDS | Does Not Receive the OUD-CDS
Number analyzed (Participants) | 5538 | 5353
dollars | -1971 [-3021 to 920] | -903 [-2143 to 337]
Statistical Analysis 1: Comparison: Receives OUD-CDS vs Does Not Receive the OUD-CDS; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Net) = -1068 — Generalized estimating equation comparing post- to pre-index costs in OUD-CDS vs. Usual Care, adjusted for site and balancing factors

8. Secondary Outcome: All-cause Mortality Per 100 Patient-years.
Time Frame: index visit through one year post-index, inclusive
Measure: Number (95% Confidence Interval); unit: events per 100 patient-years
Arm/Group | Receives OUD-CDS | Does Not Receive the OUD-CDS
Number analyzed (Participants) | 5538 | 5353
events per 100 patient-years | 2.79 [2.33 to 3.35] | 2.64 [2.23 to 3.12]
Statistical Analysis 1: Comparison: Receives OUD-CDS vs Does Not Receive the OUD-CDS; Test type: Superiority; p < 0.05, Mixed Models Analysis; Odds Ratio (OR) = 1.06

9. Secondary Outcome: Overdoses Per 100 Patient-years.
Time Frame: as for outcome 5
Measure: Number (95% Confidence Interval); unit: events per 100 patient-years
Arm/Group | Receives OUD-CDS | Does Not Receive the OUD-CDS
Number analyzed (Participants) | 5538 | 5353
events per 100 patient-years
  pre-index | 4.51 [3.69 to 5.52] | 5.32 [4.21 to 6.73]
  post-index | 3.13 [2.57 to 3.83] | 3.42 [2.73 to 4.28]
Statistical Analysis 1: Comparison: Receives OUD-CDS vs Does Not Receive the OUD-CDS; Test type: Superiority; p < 0.05, Mixed Models Analysis; Risk Ratio (RR) = 1.08 — Generalized estimating equation comparing post- to pre-index rates in OUD-CDS vs. Usual Care, adjusted for site and balancing factors

ADVERSE EVENTS:
Time Frame: pre: one year through one day prior to the index visit; post: index visit through December 31, 2023 or date of death, whichever was first, up to 33 months
Description: The safety population included all patients who had an index visit during the accrual period. Patients who were on research exclusion lists, and thus excluded from the primary study analyses, were retained for safety analyses. Safety events were monitored via passive surveillance of EHR and healthcare claims data.
Arm/Group | Receives OUD-CDS | Does Not Receive the OUD-CDS
All-Cause Mortality (participants affected / at risk) | 270/5688 | 268/5509
Serious Adverse Events (participants affected / at risk) | 3740/5688 | 3752/5509
Other Adverse Events (participants affected / at risk) | 375/5688 | 413/5509
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Receives OUD-CDS (N=5688) | Does Not Receive the OUD-CDS (N=5509)
Emergency Visits, pre-index (General disorders) | 2591 (7519) | 2578 (7723) — Emergency Department visits were counted between one year through one day prior to the index visit.
Emergency Visits, post-index (General disorders) | 2643 (9560) | 2737 (10443) — Emergency Visits were counted between the index visit and December 31, 2023 or date of death, whichever was first.
Hospitalizations, pre-index (General disorders) | 1198 (2260) | 1221 (2290) — Hospitalizations were counted between one year through one day prior to the index visit.
Hospitalizations, post-index (General disorders) | 1248 (2784) | 1285 (3000) — Hospitalizations were counted between the index visit and December 31, 2023 or date of death, whichever was first
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Receives OUD-CDS (N=5688) | Does Not Receive the OUD-CDS (N=5509)
Overdoses, pre-index (Injury, poisoning and procedural complications) | 204 (277) | 228 (326) — Overdoses were counted between one year through one day prior to the index visit.
Overdoses, post-index (Injury, poisoning and procedural complications) | 213 (326) | 225 (342) — Overdoses were counted between the index visit and December 31, 2023 or date of death, whichever was first

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI(s) should present the study primary outcome and other results to the participating sites as soon after the analyses are completed, to ensure that participating sites have a chance to comment on the results and conclusions of the trial.

The PI(s) should present primary outcome results to the Steering Committee, NIDA leadership, and the DSMB prior to publication or presentations to the public.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT04198428/Prot_SAP_001.pdf